CLINICAL TRIAL: NCT07040241
Title: Diagnostic Yield and Safety of Probe-based COnfocaL LAser Endomicroscopy and Ultrasound-guided Pleural BiOpsy in Diagnosing Patients With Unknown pleuRAl Effusion: a Protocol of a Multicenter, Randomized cONtrolled Trial (COLLABORATION-Ⅱ）
Brief Title: Confocal Laser Endomicroscopy Assisted Ultrasound Guided Pleural Biopsy
Acronym: Confocal laser
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Deputy Director of the Department of Pulmonary and Critical Care Medicine, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2025-COLLABERATION-Ⅱ
Record Dates: First submitted 2025-06-08; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pleural Effusion Disorder
Keywords: Pleural effusion; Confocal laser endomicroscopy; Pleural biopsy
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLE-assisted ultrasound-guided pleural biopsy (Experimental): The patients in this arm will receive the CLE-assisted ultrasound-guided pleural biopsy
  Interventions: Procedure: Confocoal laser endomicroscopy-assisted ultrasound-guided pleural biopsy
- Ultrasound-guided pleural biopsy (Placebo Comparator): The patients in this arm will receive the ultrasound-guided pleural biopsy
  Interventions: Procedure: Ultrasound-guided pleural biopsy

INTERVENTIONS:
Procedure: Confocoal laser endomicroscopy-assisted ultrasound-guided pleural biopsy — Using the probe-based confocal laser endomicroscopy to detect the pleural, and ensure the biopsy location. Then, use the pleural biopsy tool to complete the pleural biopsy. The whole procession will under the ultrasound guidance.
  Other Names: CLE-assisted ultrasound-guided pleural biopsy
  Arms: CLE-assisted ultrasound-guided pleural biopsy
Procedure: Ultrasound-guided pleural biopsy — Using ultrasound to detect the biopsy site and perform pleural biopsy.
  Arms: Ultrasound-guided pleural biopsy

SUMMARY:
This study aimed to evaluate the diagnostic yield and safety of confocal laser endomicroscopy and ultrasound-guided pleural biopsy in diagnosing patients with unknown pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with exudative pleural effusion of unknown origin
* Patients with negative pleural fluid cytology results
* Patients diagnosed with a probable malignant pleural effusion but without a definite diagnosis and requiring further pathological evaluation
* Patients who are fully informed of the purpose and method of the study, agree to participate in the study, and sign an informed consent form

Exclusion Criteria:

* Inability or refusal to undergo UGBx
* Patients with any contraindications for pleural biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | The day 7 after patients received CLE-assisted ultrasound-guided pleural biopsy.
  The proportion of all individuals undergoing the diagnostic procedure under evaluation in whom a specific diagnosis is established based on the consensus definition.